CLINICAL TRIAL: NCT02570659
Title: A Randomized Controlled Trial Evaluating the Effect of an Information Video in a Acute Whiplash Population
Brief Title: Investigating the Effect of an Information Video for Neck Injuries in a Emergency Department Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eric Rydman, Med dr, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Erics Whiplash RCT
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Whiplash Syndrome
Keywords: WAD; Whiplash; Information Video
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Information Folder (No Intervention): A folder with advise and exercises used by physiotherapeutic clinic of Södersjukhuset Hospital (Treatment as usual)
- Information Video (Experimental): A multiprofessional information video
  Interventions: Behavioral: Information Video

INTERVENTIONS:
Behavioral: Information Video — A 14 minutes intervention video explaining the mechanism of the injury from cross-professional point of view and physiotherapeutic advise
  Arms: Information Video

SUMMARY:
A randomized controlled trial (RCT) to investigate the effect of a information video, consisting of a multiprofessional team, on patients with acute Whiplash Associated Disorder (WAD).

DETAILED DESCRIPTION:
Patients seeking medical care at Södersjukhuset Hospital, Sweden, after a motor vehicle accident resulting in neck trauma are offered to be included in the study. Inclusion criterias involve spine fractures, need for in house care, <18<65 years of age and low knowledge of the Swedish language.

A randomization is performed with two arms, one being "treatment as usual" i.e. an information folder with physiotherapeutic exercises, the other one being the Information Video.

The patients are contacted per telephone and a questionnaire with baseline data is sent via e-mail within a week after the accident. They also receive a link to the websites with the information.

The follow up time is 6 months and after that the patients receive a new questionnaire with questions regarding neck-specific status (WDQ), health related quality of life (SF-12) and pain.

The primary outcome is level of pain (NRS)

ELIGIBILITY:
Inclusion Criteria:

* Knowledge of the swedish language
* Traffic injury with neck pain

Exclusion Criteria:

* Fractures
* In house care needed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 months
  Self reported pain the last three days (NRS)

SECONDARY OUTCOMES:
Whiplash Disability Questionnaire (WDQ) | 6 months
SF-12 | 6 months
  Health related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Eric Rydman, Stockholm, Sweden